CLINICAL TRIAL: NCT04322500
Title: Intestinal Microbiota: a New Target for Chalaziosis Treatment in Children
Brief Title: Probiotics for Chalaziosis Treatment in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Molise (Other)
Responsible Party: Principal Investigator, Ciro Costagliola, Full Professor in Ophthalmology, University of Molise
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 07/2019
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Chalazion
Keywords: microbiome/microbiota; probiotics; chalaziosis; children
MeSH Terms: conditions — Chalazion | interventions — Probiotics; Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Prospective comparative pilot study with two groups randomly divided
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: conservative (Other): conservative treatment
  Interventions: Other: conservative treatment
- Group B: probiotics (Experimental): in addition to the conservative treatment they receive a probiotics mixture (Streptococcus thermophilus ST10, Lactococcus lactis LLCO2 and Lactobacillus delbrueckii subsp. bulgaricus LDB01)
  Interventions: Dietary Supplement: probiotics; Other: conservative treatment

INTERVENTIONS:
Dietary Supplement: probiotics — use specific probiotics in addiction to conservative treatment to modify the intestinal microbiome to ameliorate the clinical course of chalaziosis in children by re-establishing intestinal and immune homeostasis
  Arms: Group B: probiotics
Other: conservative treatment — lid hygiene, warm compression, and dexamethasone/tobramycin ointment for at least 20 days

SUMMARY:
There is growing evidence encouraging the use of probiotics in many conditions in children. The aim of the investigator's study is to define the possible beneficial impact of probiotics on paediatric patients affected by chalaziosis.

DETAILED DESCRIPTION:
Prospective comparative pilot study on 26 children suffering from chalaziosis. They will be randomly divided in two groups. One group will receive conservative treatment and the other one will receive conservative treatment and a daily supplementation of probiotics. All patients will be evaluated at 2-week intervals for 3 months. If the lesion will not disappear or decrease in size to 1 mm or less in diameter on subsequent visits, the same procedure will be repeated for another 3-months cycle. The follow up periods extend from 3 to 6 months according to the results.

ELIGIBILITY:
Inclusion Criteria:

* paediatric patients
* presence of one or more eyelid mass lesions (history of rapid onset of painful inflamed mass that had reached a stationary size for more than 2 months)

Exclusion Criteria:

* eyelid infection
* chalazion duration < 1 month
* nonpalpable chalazion
* suspicion of malignancy

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Costagliola, Full Professor, Principal Investigator — University of Molise
Locations (1):
- University of Molise, Campobasso, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerry RG, Patra JK, Gouda S, Park Y, Shin HS, Das G. Benefaction of probiotics for human health: A review. J Food Drug Anal. 2018 Jul;26(3):927-939. doi: 10.1016/j.jfda.2018.01.002. Epub 2018 Feb 2. PMID 29976412
- [Background] McLean MH, Dieguez D Jr, Miller LM, Young HA. Does the microbiota play a role in the pathogenesis of autoimmune diseases? Gut. 2015 Feb;64(2):332-41. doi: 10.1136/gutjnl-2014-308514. Epub 2014 Nov 21. PMID 25416067
- [Background] Scher JU, Littman DR, Abramson SB. Microbiome in Inflammatory Arthritis and Human Rheumatic Diseases. Arthritis Rheumatol. 2016 Jan;68(1):35-45. doi: 10.1002/art.39259. No abstract available. PMID 26331579
- [Background] Ochoa-Reparaz J, Kasper LH. The influence of gut-derived CD39 regulatory T cells in CNS demyelinating disease. Transl Res. 2017 Jan;179:126-138. doi: 10.1016/j.trsl.2016.07.016. Epub 2016 Jul 28. PMID 27519147
- [Background] Kalyana Chakravarthy S, Jayasudha R, Sai Prashanthi G, Ali MH, Sharma S, Tyagi M, Shivaji S. Dysbiosis in the Gut Bacterial Microbiome of Patients with Uveitis, an Inflammatory Disease of the Eye. Indian J Microbiol. 2018 Dec;58(4):457-469. doi: 10.1007/s12088-018-0746-9. Epub 2018 Jun 4. PMID 30262956
- [Background] Iovieno A, Lambiase A, Sacchetti M, Stampachiacchiere B, Micera A, Bonini S. Preliminary evidence of the efficacy of probiotic eye-drop treatment in patients with vernal keratoconjunctivitis. Graefes Arch Clin Exp Ophthalmol. 2008 Mar;246(3):435-41. doi: 10.1007/s00417-007-0682-6. Epub 2007 Nov 27. PMID 18040708
- [Background] Tavakoli A, Flanagan JL. The Case for a More Holistic Approach to Dry Eye Disease: Is It Time to Move beyond Antibiotics? Antibiotics (Basel). 2019 Jun 30;8(3):88. doi: 10.3390/antibiotics8030088. PMID 31262073
- [Background] Lin P. The role of the intestinal microbiome in ocular inflammatory disease. Curr Opin Ophthalmol. 2018 May;29(3):261-266. doi: 10.1097/ICU.0000000000000465. PMID 29538183
- [Background] Baim AD, Movahedan A, Farooq AV, Skondra D. The microbiome and ophthalmic disease. Exp Biol Med (Maywood). 2019 Apr;244(6):419-429. doi: 10.1177/1535370218813616. Epub 2018 Nov 21. PMID 30463439
- [Background] Kugadas A, Gadjeva M. Impact of Microbiome on Ocular Health. Ocul Surf. 2016 Jul;14(3):342-9. doi: 10.1016/j.jtos.2016.04.004. Epub 2016 May 14. PMID 27189865
- [Background] Lin P. Importance of the intestinal microbiota in ocular inflammatory diseases: A review. Clin Exp Ophthalmol. 2019 Apr;47(3):418-422. doi: 10.1111/ceo.13493. Epub 2019 Mar 25. PMID 30834680
- [Background] Sansotta N, Peroni DG, Romano S, Rugiano A, Vuilleumier P, Baviera G; Italian Society of Pediatric Allergy, Immunology (SIAIP), Microbiota Committee, Italy. The good bugs: the use of probiotics in pediatrics. Curr Opin Pediatr. 2019 Oct;31(5):661-669. doi: 10.1097/MOP.0000000000000808. PMID 31356353
- [Background] Sklar BA, Gervasio KA, Leng S, Ghosh A, Chari A, Wu AY. Management and outcomes of proteasome inhibitor associated chalazia and blepharitis: a case series. BMC Ophthalmol. 2019 May 14;19(1):110. doi: 10.1186/s12886-019-1118-x. PMID 31088416
- [Background] Malekahmadi M, Farrahi F, Tajdini A. Serum Vitamin A Levels in Patients with Chalazion. Med Hypothesis Discov Innov Ophthalmol. 2017 Fall;6(3):63-66. PMID 29392144
- [Background] Yam JC, Tang BS, Chan TM, Cheng AC. Ocular demodicidosis as a risk factor of adult recurrent chalazion. Eur J Ophthalmol. 2014 Mar-Apr;24(2):159-63. doi: 10.5301/ejo.5000341. Epub 2013 Jul 16. PMID 23873491
- [Background] Lu LJ, Liu J. Human Microbiota and Ophthalmic Disease. Yale J Biol Med. 2016 Sep 30;89(3):325-330. eCollection 2016 Sep. PMID 27698616
- See also: probiotics definition — http://fao.org/3/a-a0512e.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Group B: Probiotics: in addition to the conservative treatment they receive a probiotics mixture (ST10, LLCO2 and LDB01)
  probiotics: use specific probiotics in addiction to conservative treatment to modify the intestinal microbiome to ameliorate the clinical course of chalaziosis in children by re-establishing intestinal and immune homeostasis
  conservative treatment: lid hygiene, warm compression, and dexamethasone/tobramycin ointment for at least 20 days
Period: Overall Study
Arm/Group | Group A: Conservative | Group B: Probiotics
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Conservative | Group B: Probiotics | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (1.2) | 8.6 (1.9) | 8.3 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Time Taken for a Complete Resolution of the Chalaziosis
Description: change in the time taken for complete resolution of chalaziosis (complete disappearance of the eyelid mass lesions)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A: Conservative | Group B: Probiotics
Number analyzed (Participants) | 13 | 13
days | 51.2 (12.4) | 28.4 (10.8)

2. Primary Outcome: Number of Recurrences
Description: complete ophthalmological evaluation was done weekly during the first month and then monthly in order to evaluate possible recurrences (presence of a new eyelid mass lesion)
Time Frame: 3 months
Measure: Number; unit: recurreces
Arm/Group | Group A: Conservative | Group B: Probiotics
Number analyzed (Participants) | 13 | 13
recurreces | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group A: Conservative | Group B: Probiotics
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Further studies are needed to confirm this first pilot trial (larger cohort, ocular and gut microbiome analysis).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04322500/Prot_SAP_000.pdf